CLINICAL TRIAL: NCT04397367
Title: Low Dose Ruxolitinib in Combination With Methylprednisolone 1mg/kg as Initial Therapy for Acute Graft-Versus-Host Disease
Brief Title: Low Dose Ruxolitinib in Combination With Methylprednisolone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: S-2019-177-01
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: aGVHD; Stem Cell Transplant Complications
MeSH Terms: interventions — ruxolitinib; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ruxolitinib10 mg twice a day combined with Corticosteroids (Experimental): Newly diagnosed acute GVHD patients started therapy with methylprednisolone of 1 mg/kg/day after diagnosis. Ruxolitinib was administered at a median of 2 days after the use of methylprednisolone. Participants began oral administration of ruxolitinib at 10 mg twice a day. Ruxolitinib was subsequently tapered due to the resolution of acute GVHD after three months of therapy. A dose-tapering schedule that would discontinue ruxolitinib in three months was recommended.
  Interventions: Drug: Ruxolitinib 10 mg twice a day combined with Corticosteroids
- Ruxolitinib5 mg twice a day combined with Corticosteroids (Experimental): Newly diagnosed acute GVHD patients started therapy with methylprednisolone of 1 mg/kg/day after diagnosis. Ruxolitinib was administered at a median of 2 days after the use of methylprednisolone. Participants began oral administration of ruxolitinib at 5 mg twice a day. Ruxolitinib was subsequently tapered due to the resolution of acute GVHD after three months of therapy. A dose-tapering schedule that would discontinue ruxolitinib in three months was recommended.
  Interventions: Drug: Ruxolitinib 5 mg twice a day combined with Corticosteroids
- Ruxolitinib5 mg once a day combined with Corticosteroids (Experimental): Newly diagnosed acute GVHD patients started therapy with methylprednisolone of 1 mg/kg/day after diagnosis. Ruxolitinib was administered at a median of 2 days after the use of methylprednisolone. Participants began oral administration of ruxolitinib at 5mg once a day. Ruxolitinib was subsequently tapered due to the resolution of acute GVHD after three months of therapy. A dose-tapering schedule that would discontinue ruxolitinib in three months was recommended.
  Interventions: Drug: Ruxolitinib 5 mg once a day combined with Corticosteroids
- Ruxolitinib 2.5 mg twice a day combined with Corticosteroids (Experimental): Newly diagnosed acute GVHD patients started therapy with methylprednisolone of 1 mg/kg/day after diagnosis. Ruxolitinib was administered at a median of 2 days after the use of methylprednisolone. Participants began oral administration of ruxolitinib at 2.5 mg once a day. Ruxolitinib was subsequently tapered due to the resolution of acute GVHD after three months of therapy. A dose-tapering schedule that would discontinue ruxolitinib in three months was recommended.
  Interventions: Drug: Ruxolitinib 2.5 mg once a day combined with Corticosteroids

INTERVENTIONS:
Drug: Ruxolitinib 10 mg twice a day combined with Corticosteroids — Newly diagnosed acute GVHD patients started therapy with methylprednisolone of 1 mg/kg/day after diagnosis. Ruxolitinib was administered at a median of 2 days after the use of methylprednisolone. Participants began oral administration of ruxolitinib at 10 mg twice a day. Ruxolitinib was subsequently tapered due to the resolution of acute GVHD after three months of therapy. A dose-tapering schedule that would discontinue ruxolitinib in three months was recommended.
  Other Names: ruxolitinib 10 mg twice a day
  Arms: Ruxolitinib10 mg twice a day combined with Corticosteroids
Drug: Ruxolitinib 5 mg twice a day combined with Corticosteroids — Newly diagnosed acute GVHD patients started therapy with methylprednisolone of 1 mg/kg/day after diagnosis. Ruxolitinib was administered at a median of 2 days after the use of methylprednisolone. Participants began oral administration of ruxolitinib at 5 mg twice a day. Ruxolitinib was subsequently tapered due to the resolution of acute GVHD after three months of therapy. A dose-tapering schedule that would discontinue ruxolitinib in three months was recommended.
  Other Names: ruxolitinib 5 mg twice a day
  Arms: Ruxolitinib5 mg twice a day combined with Corticosteroids
Drug: Ruxolitinib 5 mg once a day combined with Corticosteroids — Newly diagnosed acute GVHD patients started therapy with methylprednisolone of 1 mg/kg/day after diagnosis. Ruxolitinib was administered at a median of 2 days after the use of methylprednisolone. Participants began oral administration of ruxolitinib at 5 mg once a day. Ruxolitinib was subsequently tapered due to the resolution of acute GVHD after three months of therapy. A dose-tapering schedule that would discontinue ruxolitinib in three months was recommended.
  Other Names: Ruxolitinib 5 mg once a day
  Arms: Ruxolitinib5 mg once a day combined with Corticosteroids
Drug: Ruxolitinib 2.5 mg once a day combined with Corticosteroids — Newly diagnosed acute GVHD patients started therapy with methylprednisolone of 1 mg/kg/day after diagnosis. Ruxolitinib was administered at a median of 2 days after the use of methylprednisolone. Participants began oral administration of ruxolitinib at 2.5 mg once a day. Ruxolitinib was subsequently tapered due to the resolution of acute GVHD after three months of therapy. A dose-tapering schedule that would discontinue ruxolitinib in three months was recommended.
  Other Names: Ruxolitinib 2.5 mg once a day
  Arms: Ruxolitinib 2.5 mg twice a day combined with Corticosteroids

SUMMARY:
This study is to determine the efficacy and safety of combined Low dose Ruxolitinib With Methylprednisone as Initial Therapy for the aGVHD(acute graft-versus-host disease )

DETAILED DESCRIPTION:
Corticosteroid is used as a first-line treatment for acute GVHD. However, it is effective in only about half of patients. In this prospective study, the investigators prospectively combined low dose ruxolitinib and 1mg/kg methylprednisolone in the initial treatment of acute GVHD. In order to effectively control GVHD without exposing acute GVHD patients to more intense and prolonged immunosuppression, we used ruxolitinib (20mg/day, 10mg/day, 5mg/day, 2.5mg/day) combined with 1mg/kg methylprednisolone. To ally steroid-related complications, we decreased steroid exposure time (39 days) and cumulative methylprednisolone doses (15.4 mg/kg) to spare the associated toxicity of glucocorticoid therapy.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with hematological diseases.
2. Have undergone first allogeneic hematopoietic stem cell transplantation (allo-HSCT) from any donor source using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies.
3. new onset of grade II~IV aGVHD or high risk aGVHD [based on suppression of tumorigenicity 2 (also ST2), Regenerating Islet Derived Protein 3 Alpha (also REG3a), experimental objects) within 100 days post-transplantation.

Exclusion Criteria:

1. recipients of second allogeneic stem cell transplant.
2. acute GVHD induced by donor lymphocyte infusion, interferon.
3. received first line aGVHD treatment before enrollment.
4. overlap GVHD syndrome.
5. pregnant or breast-feeding women.
6. absolute neutrophil count (ANC) <0.5×10e9/L or platelet count (PLT) < 20×10e9/L
7. Serum creatinine > 2.0 mg/dL or creatinine clearance < 40 mL/min measured or calculated by Cockroft-Gault equation.
8. uncontrolled infection
9. human immunodeficiency virus infection
10. active hepatitis b virus, hepatitis C virus infection and need antivirus treatment.
11. Subjects with evidence of relapsed primary disease, or subjects who have been treated for relapse after the allo-HSCT was performed, or graft rejection.
12. allergic history to Janus kinase inhibitors.
13. Severe organ dysfunction unrelated to underlying GVHD, including:

    Cholestatic disorders or unresolved veno-occlusive disease of the liver (defined as persistent bilirubin abnormalities not attributable to GVHD and ongoing organ dysfunction). Clinically significant or uncontrolled cardiac disease including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic support, or arrhythmia that requires therapy. Clinically significant respiratory disease that requires mechanical ventilation support or 50% oxygen.
14. Received Janus kinase inhibitor therapy after allo-HSCT for any indication.
15. Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
complete remission rate of acute GVHD 28 days after enrollment. | Day 28 after treatment
  Defined as the proportion of participants demonstrating a complete response (CR), or partial response (PR) of acute GVHD

SECONDARY OUTCOMES:
the incidence of relapsed acute GVHD | Day 90 after treatment
  Defined as the proportion of participants whose improved acute GVHD.
Six-month duration of response | Six-month after treatment
  Defined as the time from first response until graft-versus-host disease (GVHD) progression or death. Duration of response will be assessed when all participants who are still on study complete the Day 180 visit.
Duration of response | Day 90 after treatment
  Defined as the time from first response until GVHD progression or death, when all participants who are still on study complete the Day 90 visit.
Nonrelapse mortality (NRM) | 6 months after treatment
  Defined as the proportion of subjects who died due to causes other than malignancy relapse.
Relapse rate | 2 years after treatment
  Defined as the proportion of participants whose underlying malignancy relapsed.

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dou LP, Li HH, Wang L, Li F, Huang WR, Yu L, Liu DH. Efficacy and Safety of Unmanipulated Haploidentical Related Donor Allogeneic Peripheral Blood Stem Cell Transplantation in Patients with Relapsed/Refractory Acute Myeloid Leukemia. Chin Med J (Engl). 2018 Apr 5;131(7):790-798. doi: 10.4103/0366-6999.228243. PMID 29578122
- [Background] Sandmaier BM, Kornblit B, Storer BE, Olesen G, Maris MB, Langston AA, Gutman JA, Petersen SL, Chauncey TR, Bethge WA, Pulsipher MA, Woolfrey AE, Mielcarek M, Martin PJ, Appelbaum FR, Flowers MED, Maloney DG, Storb R. Addition of sirolimus to standard cyclosporine plus mycophenolate mofetil-based graft-versus-host disease prophylaxis for patients after unrelated non-myeloablative haemopoietic stem cell transplantation: a multicentre, randomised, phase 3 trial. Lancet Haematol. 2019 Aug;6(8):e409-e418. doi: 10.1016/S2352-3026(19)30088-2. Epub 2019 Jun 24. PMID 31248843
- [Result] Ruutu T, Gratwohl A, Niederwieser D, de Witte T, van der Werf S, van Biezen A, Mohty M, Kroger N, Rambaldi A, McGrath E, Sureda A, Basak G, Greinix H, Duarte RF. The EBMT-ELN working group recommendations on the prophylaxis and treatment of GvHD: a change-control analysis. Bone Marrow Transplant. 2017 Mar;52(3):357-362. doi: 10.1038/bmt.2016.298. Epub 2016 Nov 28. PMID 27892949
- [Result] Akahoshi Y, Igarashi A, Fukuda T, Uchida N, Tanaka M, Ozawa Y, Kanda Y, Onizuka M, Ichinohe T, Tanaka J, Atsuta Y, Kako S; Adult Acute Lymphoblastic Leukemia Working Group of the Japan Society for Hematopoietic Cell Transplantation. Impact of graft-versus-host disease and graft-versus-leukemia effect based on minimal residual disease in Philadelphia chromosome-positive acute lymphoblastic leukemia. Br J Haematol. 2020 Jul;190(1):84-92. doi: 10.1111/bjh.16540. Epub 2020 Mar 2. PMID 32119132
- [Result] Yeshurun M, Weisdorf D, Rowe JM, Tallman MS, Zhang MJ, Wang HL, Saber W, de Lima M, Sandmaier BM, Uy G, Kamble RT, Cairo MS, Cooper BW, Cahn JY, Ganguly S, Camitta B, Verdonck LF, Dandoy C, Diaz MA, Savani BN, George B, Liesveld J, McGuirk J, Byrne M, Grunwald MR, Drobyski WR, Pulsipher MA, Abdel-Azim H, Prestidge T, Wieduwilt MJ, Martino R, Norkin M, Beitinjaneh A, Seo S, Nishihori T, Wirk B, Frangoul H, Bashey A, Mori S, Marks DI, Bachanova V. The impact of the graft-versus-leukemia effect on survival in acute lymphoblastic leukemia. Blood Adv. 2019 Feb 26;3(4):670-680. doi: 10.1182/bloodadvances.2018027003. PMID 30808685
- [Result] Zeiser R, Burchert A, Lengerke C, Verbeek M, Maas-Bauer K, Metzelder SK, Spoerl S, Ditschkowski M, Ecsedi M, Sockel K, Ayuk F, Ajib S, de Fontbrune FS, Na IK, Penter L, Holtick U, Wolf D, Schuler E, Meyer E, Apostolova P, Bertz H, Marks R, Lubbert M, Wasch R, Scheid C, Stolzel F, Ordemann R, Bug G, Kobbe G, Negrin R, Brune M, Spyridonidis A, Schmitt-Graff A, van der Velden W, Huls G, Mielke S, Grigoleit GU, Kuball J, Flynn R, Ihorst G, Du J, Blazar BR, Arnold R, Kroger N, Passweg J, Halter J, Socie G, Beelen D, Peschel C, Neubauer A, Finke J, Duyster J, von Bubnoff N. Ruxolitinib in corticosteroid-refractory graft-versus-host disease after allogeneic stem cell transplantation: a multicenter survey. Leukemia. 2015 Oct;29(10):2062-8. doi: 10.1038/leu.2015.212. Epub 2015 Jul 31. PMID 26228813
- [Result] Walker I, Panzarella T, Couban S, Couture F, Devins G, Elemary M, Gallagher G, Kerr H, Kuruvilla J, Lee SJ, Moore J, Nevill T, Popradi G, Roy J, Schultz KR, Szwajcer D, Toze C, Foley R; Cell Therapy Transplant Canada. Addition of anti-thymocyte globulin to standard graft-versus-host disease prophylaxis versus standard treatment alone in patients with haematological malignancies undergoing transplantation from unrelated donors: final analysis of a randomised, open-label, multicentre, phase 3 trial. Lancet Haematol. 2020 Feb;7(2):e100-e111. doi: 10.1016/S2352-3026(19)30220-0. Epub 2020 Jan 17. PMID 31958417